CLINICAL TRIAL: NCT05490342
Title: Evaluation of SARS-CoV-2 Antibody Response After Vaccination in Liver Transplant Recipients Who Undergo Tailored Immunosuppression Therapy
Brief Title: Effect of SARS-CoV-2 Vaccination in Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Tommaso Maria Manzia, Associate Professor, University of Rome Tor Vergata
Other Study IDs: sperimentazioni PTV 71.22
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2 Vaccination; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tacrolimus-based immunosuppresion: The TAC-based group will include any patient on tacrolimus monotherapy and patients taking multiple IS medications with blood tacrolimus levels > 5 ng/mL
  Interventions: Diagnostic Test: Immunoassay, by ECLIA, for the quantitative in vitro determination of antibodies (including IgG) to the SARS - CoV - 2 spike protein (S) anti-RBD (receptor-binding domain) in serum and plasma samples.
- NON-tacrolimus-based immunosuppresion: The NON-TAC-based group will include any patient on TAC-free therapy and patient taking multiple IS medications with blood tacrolimus levels < 5 ng/mL
  Interventions: Diagnostic Test: Immunoassay, by ECLIA, for the quantitative in vitro determination of antibodies (including IgG) to the SARS - CoV - 2 spike protein (S) anti-RBD (receptor-binding domain) in serum and plasma samples.

INTERVENTIONS:
Diagnostic Test: Immunoassay, by ECLIA, for the quantitative in vitro determination of antibodies (including IgG) to the SARS - CoV - 2 spike protein (S) anti-RBD (receptor-binding domain) in serum and plasma samples. — Blood test to value the antibody response to vaccination

SUMMARY:
To investigate the variations in the humoral response to vaccines for the prevention of COVID-19 in liver transplant patients based on the type of immunosuppressive therapy adopted (tacrolimus based vs no-tacrolimus based) and immunosuppressive blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplanted patients >18 years of age.
* Patients who underwent liver transplantation between 01/2015 to 12/2021.
* Patients who underwent liver transplantation at "Policlinico Tor Vergata, Rome, Italy".
* Patients who have had three doses of a vaccine for the prevention of COVID-19.
* Patients who have had three doses of a SARS-CoV-2 vaccine and who have contracted SARS-CoV-2 infection.

Exclusion Criteria:

* Patients who have more or less than three dose of a vaccine for the prevention of COVID-19
* Patients not vaccinated for prevention of SARS-CoV-2 infection.
* Patients who have had three doses of a vaccine for the prevention of COVID-19 prior to liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant recipients who underwent SARS-CoV-2 vaccination (3 doses)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of positive antibody titer | Between 30 and 120 ± 15 days after the completion of the vaccination cycle
  > 0.8 U/mL

SECONDARY OUTCOMES:
Rate of highly protective antibody titer | Between 30 and 120 ± 15 days after the completion of the vaccination cycle
  >100 BAU/mL
Median antibody titer absolute value | Between 30 and 120 ± 15 days after the completion of the vaccination cycle
  BAU/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata, Roma, Italy

IPD SHARING:
Plan to Share IPD: No